CLINICAL TRIAL: NCT02776553
Title: A Physical Activity Program in End-stage Liver Disease: Pilot Study Assessing Changes in Physical Fitness, Sarcopenia, and the Metabolic Profile
Brief Title: A Physical Activity Program in End-state Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 203659
Record Dates: First submitted 2016-05-13; First posted 2016-05-18 (Estimated); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: End-stage Liver Disease (ESLD); Liver Transplant; Sarcopenia; Poor Physical Fitness; Cirrhosis; Portal Hypertension
MeSH Terms: conditions — End Stage Liver Disease; Sarcopenia; Fibrosis; Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (physical training program) (Experimental): physical activity + behavioral therapy + nutritional intervention
  Interventions: Other: Nutritional consultation; Behavioral: Physical training program; Behavioral: Behavioral modification therapy
- Control (Active Comparator): nutritional intervention
  Interventions: Other: Nutritional consultation

INTERVENTIONS:
Other: Nutritional consultation — Dietary advice will be provided at the beginning of the study and individually tailored to the participant's usual eating habits plus amino acid supplement including 10 grams of branched-chain amino acids
Behavioral: Physical training program — Physical activity prescription will target ≥10,000 steps/day, taking into account all activities performed throughout the day, although the increment in activity should be no less than 3000 steps/day above the baseline.
  Arms: Active (physical training program)
Behavioral: Behavioral modification therapy — The behavior modification theory will be applied in the form of a structured set of cues and questions between investigator and participant at each visit in order to provide individually tailored counseling to enhance internal motivation and facilitate behavior change toward physical activity and dietary improvement that are adaptable to each participant's usual habits.
  Arms: Active (physical training program)

SUMMARY:
The primary aim of this study is to improve both physical fitness and sarcopenia of patients with ESLD who are potentially eligible for liver transplantation through a 12-week physical training program. Secondary aims will focus on changes in anthropometrics, body composition, quality of life, and metabolic profile. This is a randomized clinical trial including 50 patients, with half allocated to the active group (physical training program) and half to standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 70.
* Cirrhosis, any cause, defined as:

  * Biopsy-proven.
  * Two or more of the following: albumin <3.5 g/dL, International Normalized Ration (INR) >1.3, radiologic or endoscopic evidence of portal hypertension.
* Creatinine <2.0 mg/dL.
* Physiologic Model for End Stage Liver Disease (MELD) ≥10.
* Decompensated cirrhosis with active or history of variceal bleeding, ascites, hepatic encephalopathy, or jaundice.
* Potential transplant candidate as per UAMS criteria

Exclusion Criteria:

* Large gastric or esophageal varices with contraindication to use beta-blockers.
* Persistent hepatic encephalopathy grades 2-4.
* Prior diagnosis of hepatocellular carcinoma, or hepatic hydrothorax (with prior repeated thoracocentesis).
* Cirrhotic cardiomyopathy or congestive heart failure, pulmonary vascular complications, known active coronary artery disease, syncope, and cardiac dysrhythmias.
* Physical impediment to perform a cardiorespiratory fitness test.
* Use of implantable defibrillator or a pacemaker.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2020-05 (Actual); Study Completion 2020-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andres Duarte-Rojo, MD, Principal Investigator — University of Arkansas Medical Sciences
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 227 Subjects were recruited from the UAMS liver transplant clinic. 207 were excluded for meeting exclusion criteria.
Period: Overall Study
Arm/Group | Active (Physical Training Program) | Control
Started | 9 (One subject was eliminated for repeated hospitalizations.) | 8 (Two subjects were eliminated for repeated hospitalizations.)
Completed | 6 | 5
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — got liver transplant | 1 | 2
Not completed — had other surgery | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active (Physical Training Program) | Control | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (7) | 54 (11) | 55 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 8 | 7 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 8 | 7 | 15
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Etiology of cirrhosis-NASH/cryptogenic [Count of Participants; unit: Participants] | 1 | 4 | 5
Etiology of cirrhosis-Hepatitis C [Count of Participants; unit: Participants] | 3 | 2 | 5
Etiology of cirrhosis-Alcoholic [Count of Participants; unit: Participants] | 4 | 0 | 4
Etiology of cirrhosis-Cholestatic [Count of Participants; unit: Participants] | 1 | 2 | 3
Weight [Mean (Standard Deviation); unit: kilograms] | 92 (21) | 89 (14) | 91 (18)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31 (8) | 29 (4) | 30 (6)
Diabetes Mellitus [Count of Participants; unit: Participants] | 4 | 1 | 5
Hypertension [Count of Participants; unit: Participants] | 1 | 2 | 3
Use of beta-blocker [Count of Participants; unit: Participants] | 1 | 2 | 3
Esophageal varices [Count of Participants; unit: Participants] | 5 | 7 | 12
Prior variceal bleeding [Count of Participants; unit: Participants] | 1 | 1 | 2
Ascites [Count of Participants; unit: Participants] | 7 | 6 | 13
Large volume paracentesis [Count of Participants; unit: Participants] | 3 | 1 | 4
Hepatic encephalopathy [Count of Participants; unit: Participants] | 9 | 8 | 17
Child-Turcotte-Pugh Score [median (range)] [Median (Full Range); unit: units on a scale] — This clinical score is an indicator of severity of liver disease. It is derived from 5 clinical domains: hepatic encephalopathy, ascites, INR (international normalized ratio) or prothrombin time, serum albumin, and total bilirubin. In each domain, a score is given from 1 (best health) to 3 (worst health); therefor the total possible range is 5-15 with higher scores indicative of worse liver disease.
  units on a scale | 9 [7 to 12] | 10 [8 to 13] | 9 [7 to 13]
Child-Turcotte-Pugh Class B [Count of Participants; unit: Participants] — This clinical classification is an indicator of severity of liver disease. It is derived from the total Child-Turcotte-Pugh score (range is 5-15) with higher scores indicative of worse liver disease. A total score of 7-9 is designated Class B - moderate liver disease (worse than Class A, but better than Class C).
  Participants | 7 | 4 | 11
Child-Turcotte-Pugh Class C [Count of Participants; unit: Participants] — This clinical classification is an indicator of severity of liver disease. It is derived from the total Child-Turcotte-Pugh score (range is 5-15) with higher scores indicative of worse liver disease. A total score of 10-15 is designated Class C - severe liver disease (worse than Class A and Class B).
  Participants | 2 | 4 | 6
D'Amico Stage 4 [Count of Participants; unit: Participants] — A set of clinical criteria that is used to stratify liver disease into five stages. The criteria include presence or absence of ascites, varices, and bleeding. Higher stages indicate more severe liver disease and increased risk of death.
  Participants | 8 | 7 | 15
D'Amico Stage 5 [Count of Participants; unit: Participants] — A set of clinical criteria that is used to stratify liver disease into five stages. The criteria include presence or absence of ascites, varices, and bleeding. Higher stages indicate more severe liver disease and increased risk of death.
  Participants | 1 | 1 | 2
Total bilirubin (mg/dL) [Mean (Standard Deviation); unit: mg/dL] | 2.3 (1.3) | 3.1 (1.5) | 2.7 (1.4)
ALT [Mean (Standard Deviation); unit: units per liter] | 34 (18) | 45 (16) | 39 (16)
AST [Mean (Standard Deviation); unit: units per liter] | 54 (28) | 78 (31) | 65 (29)
Albumin [Mean (Standard Deviation); unit: g/dL] | 3.1 (0.3) | 2.5 (0.6) | 2.8 (0.5)
Hemoglobin [Mean (Standard Deviation); unit: g/dL] | 12.1 (2.6) | 11.4 (2.3) | 11.7 (2.4)
Platelets [Mean (Standard Deviation); unit: thousand platelets/microliter] | 121 (74) | 112 (24) | 116 (63)
INR [Mean (Standard Deviation); unit: units on a scale] — The international normalised ratio (INR) is a laboratory measurement of how long it takes blood to form a clot. If an INR score is too low, a patient can be at risk for a blood clot. However, if the INR is too high, patients could also experience bleeding. A typical INR score ranges between 2 to 3. The "ideal" INR score can vary from patient to patient.
  units on a scale | 1.4 (0.3) | 1.7 (1.2) | 1.5 (0.4)
Creatinine [Mean (Standard Deviation); unit: mg/dL] | 0.8 (0.3) | 0.9 (0.3) | 0.9 (0.2)
Sodium [Mean (Standard Deviation); unit: mEq/L] | 135 (3) | 135 (4) | 135 (3)
MELD-sodium [Mean (Standard Deviation); unit: units on a scale] — This is primarily used to stratify patients ≥12 years old on liver transplant waiting lists. It also predicts mortality in the following scenarios: (a) after transjugular intrahepatic portosystemic shunt (TIPS), (b) cirrhotic patients undergoing non-transplantation surgical procedures, (c) acute alcoholic hepatitis, and (d) acute variceal hemorrhage. It is derived from: the frequency of dialysis, creatinine, bilirubin, sodium, and INR (international normalised ratio-an indicator of blood-clotting efficiency). The full range is 6-40, with higher numbers indicating more severe disease.
  units on a scale | 16 (4) | 19 (3) | 17 (4)

OUTCOME MEASURES:

1. Primary Outcome: Physical Fitness - VO2
Description: Peak VO2 will be obtained from cardiorespiratory stress test
Time Frame: Change from Baseline to 12 weeks after baseline
Measure: Mean (Standard Deviation); unit: mL oxygen/kg/min
Arm/Group | Active (Physical Training Program) | Control
Number analyzed (Participants) | 9 | 8
mL oxygen/kg/min | -1 (6.5) | -3 (6.5)
Statistical Analysis 1: Comparison: Active (Physical Training Program) vs Control; Test type: Superiority; p = 0.49, ANCOVA

2. Primary Outcome: Physical Fitness - Distance Walked
Description: Total distance walked during 6-minute walk test
Time Frame: Change from Baseline to 12 weeks after baseline
Measure: Mean (Full Range); unit: meters
Arm/Group | Active (Physical Training Program) | Control
Number analyzed (Participants) | 6 | 5
meters | 59.2 [-36 to 133] | -91.4 [-291 to 27]
Statistical Analysis 1: Comparison: Active (Physical Training Program) vs Control; Test type: Superiority; p = 0.03, ANCOVA

3. Primary Outcome: Sarcopenia
Description: Total thigh muscle volume (cm^3), as determined by CT-scan.
Time Frame: Change from Baseline to 12 weeks after baseline
Measure: Mean (95% Confidence Interval); unit: cubic centimeters
Arm/Group | Active (Physical Training Program) | Control
Number analyzed (Participants) | 9 | 8
cubic centimeters | -124 [-881 to 384] | -373 [-881 to 384]
Statistical Analysis 1: Comparison: Active (Physical Training Program) vs Control; Test type: Superiority; p = 0.37, ANCOVA

ADVERSE EVENTS:
Time Frame: Approximately 4 months duration per subject.
Arm/Group | Active (Physical Training Program) | Control
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/53/NCT02776553/Prot_SAP_000.pdf